CLINICAL TRIAL: NCT05835648
Title: Effect of Dietary Fiber on Anemia and Glomerular Filtration Rate in Non-dialysis Patients With Chronic Kidney Disease
Brief Title: Effect of Dietary Fiber on Non-dialysis Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Zunsong Wang, Clinical professor, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CKD-Dietary fiber
Record Dates: First submitted 2023-03-19; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Kidney Disease
Keywords: Dietary fiber; CKD; Anemia; glomerular filtration rate
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary fiber intervention group (Experimental): On the basis of daily diet, dietary fiber supplement (Nutrasumma) was given once a day, 1 strip each time, before meals, and the intervention lasted for 3 months.
  Interventions: Dietary Supplement: Nutrasumma

INTERVENTIONS:
Dietary Supplement: Nutrasumma — On the basis of daily diet, dietary fiber supplement (Nutrasumma) was given once a day, 1 strip each time, before meals, and the intervention lasted for 3 months.

SUMMARY:
The main objective of this study was to investigate the effect of dietary fiber on anemia and glomerular filtration rate in non-dialysis patients with chronic kidney disease. Participants will be randomly divided into a dietary fiber intervention group and a blank control group. The patients in the dietary fiber intervention group will have dietary fiber intake survey conducted by dietitians on the basis of basic treatment. Supplemented dietary fiber was given on the basis of daily diet, once a day, 1 piece each time, before meals, and the intervention lasted for 3 months. The blank control group was followed up without intervention. Clinical data, blood, urine and stool samples were collected at the initial diagnosis and at each follow-up site.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old;
* Clinically confirmed (history, blood creatinine, kidney B-ultrasound, laboratory examination, etc.) as stage 3-5 chronic kidney disease, endogenous creatinine clearance was < 60ml/min according to Cockcroft-Gault formula;
* Generally in good condition, have a good understanding of their own illness and physical condition, have self-awareness, and can communicate well with others;
* Hemoglobin 100-130g/L;
* In a non-dialysis state.
* Dietary fiber intake <25g/d;
* Voluntarily join the study, understand the significance of the test and the indicators to be measured, and sign the informed consent.

Exclusion Criteria:

* Unwilling to join the study; Severe infection: fever, cough and sputum, pharyngeal pain, abdominal pain, diarrhea, carbuncle and other skin and soft tissue infection and other clinical manifestations, blood routine white blood cell count beyond the normal range (10×109/L);
* Severe cardiovascular diseases: including chronic cardiac insufficiency grade 3 or above and various arrhythmias;
* Obvious hypoproteinemia: albumin less than 30g/L;
* Corrective measures for anemia (blood transfusion, erythropoietin, HIF-PHI, iron supplement) have been applied in the past 3 months;
* Tumor evidence: certain tumors have been detected or clinical manifestations and tumor markers suggest the possibility of tumor;
* Pregnant women;
* Recent history of heavy blood loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-04-30 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in baseline hemoglobin levels at 9 months | 9 months
Changes of glomerular filtration rate at baseline at 9 months | 9 months

IPD SHARING:
Plan to Share IPD: No